CLINICAL TRIAL: NCT02315976
Title: Avaliação de episódios Agudos na Angina Pectoris crônica estável: Abordagem clínico-laboratorial do Uso do Vasodilatador Coronariano Propatilnitrato.
Brief Title: Acute Episodes in Chronic Stable Angina: Assessment of the Use of the Coronary Vasodilator Propatyl Nitrate.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundação Educacional Serra dos Órgãos (Other)
Responsible Party: Principal Investigator, Carlos Pereira Nunes, Professor of Internal Medicine, Fundação Educacional Serra dos Órgãos
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APPN 01-01-13
Record Dates: First submitted 2014-11-29; First posted 2014-12-12 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Chronic Stable Angina Pectoris
Keywords: chronic stable angina pectoris; propatyl nitrate; Seattle Angina Questionnaire
MeSH Terms: interventions — propatyl nitrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Propatyl nitrate (Experimental): Patients treated with propatyl nitrate 10mg thrice daily
  Interventions: Drug: Propatyl Nitrate

INTERVENTIONS:
Drug: Propatyl Nitrate — Propatyl nitrate 10mg administered orally, three times daily

SUMMARY:
This is an open, self-paired study of 200 patients with heart failure who have a diagnosis of chronic stable angina pectoris, who will be treated for 30 days with propatyl nitrate (10mg) . Treatment regimen is 3 sublingual tablets per day, at 8:00 AM, 2:00 PM, and 8:00 PM. The study will include three visits the patient to the study center: Pretreatment / Assessment 1, Assessment 2 after 15 days of treatment, and the Assessment 3 after 30 days of treatment. At each visit, data will be collected on the medical history, physical examination and vital signs, and evaluation of episodes of angina pectoris, as well as the laboratory evaluation of adverse events and the use of concomitant medications.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic stable angina pectoris
* Female subjects post-menopausal or not pregnant and using of contraceptives
* Signature of Informed consent document

Exclusion Criteria:

* Pregnant women or nursing patients , women of childbearing age
* Hypersensitivity or intolerance to any component of the study drug
* Angina pectoris Class IV, according to the Canadian Society of Cardiology
* Clinical diagnosis of severe anemia , glaucoma, head trauma , increased intracranial pressure, cerebral hemorrhage, acute myocardial infarction, congestive heart failure, aortic valve disease
* Recent infarction (within the last 3 months)
* Recent history (within the last 6 months)of angioplasty
* Use of these medicines within 7 days screening : sildenafil citrate and other inhibitors of phosphodiesterase-5 , adrenergic substances
* Significant alteration of any laboratory test (> 20% above or below the normal range )
* Gastric or intestinal ulcer or intestinal
* Asthma or chronic rhinitis
* Any other condition which in the opinion of the investigator, shall exclude the study of the patient.

Ages: 50 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of angina episodes | 30-day treatment period
  Number of angina episodes per patient during the 30 day treatment period

SECONDARY OUTCOMES:
Pain intensity | 30-day treatment period
  Percentage of patients with moderate (50-69mm) to severe (>70mm) pain (100mm visual analog pain scale)
Episode duration | 30-day treatment period
  Number of angina episodes lasting two or more minutes
Adverse Event - occurence | 30-day treatment period
  Number of patients presenting adverse events
Seattle Angina Questionnaire (SAQ) scales score improvements | 30-day treatment period
  Improvement greater than or equal to 30% in SAQ scales scores of physical limitation, anginal stability, treatment satisfaction, and quality of life.
Seattle Angina Questionnaire (SAQ) Score increase >30% | 30-day treatment period
  Percentage of patients with Seattle Angina Questionnaire score improvement greater than or equal to 30%

CONTACTS AND LOCATIONS:
Locations (1):
- UNIFESO, Teresópolis, Rio de Janeiro, Brazil